CLINICAL TRIAL: NCT06781424
Title: University of Central Florida Biobank for Extreme Environments, Aviation and Space Travel
Brief Title: University of Central Florida BEEAST
Status: Recruiting | Type: Observational
Sponsor: University of Central Florida (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00007332
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Biospecimen Donation; Environmental Impact
Keywords: donate; biobank; biospecimen; astronaut; pilot

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Primary Partcipant: Participants who have who travel (such as space travel) or live in extreme environments (such as Antarctica).
- Secondary Participant: Participants who have been referred adult family members (such as siblings and spouses) of primary enrollees.
- Tertiary Partcipant: Participants from the general public to serve as matching controls.

SUMMARY:
Since the inception of aerospace travel, NASA has been collecting biospecimens from professional astronauts for research. With the recent growth of civilian aerospace travelers, there is a need for biospecimen banking for civilian astronauts. This protocol addresses this gap by being a biobank for civilian astronauts, their family members (to be controls) and others who are also doing travel to extreme environments (pilots, submariners).

DETAILED DESCRIPTION:
The objective of the University of Central Florida College of Medicine's Biobank for Extreme Environments, Aviation and Space Travel (BEEAST) is to acquire, store, and distribute identifiable human biospecimens and health information for medical research purposes only. The target population are astronauts, aviators, submariners, persons living in extreme environments (such as Antarctica), and their families, and people from the general population who can serve as matching controls.

ELIGIBILITY:
Inclusion Criteria:

* Primary Enrollees: adults, ages 18 and older, and persons who travel (such as space travel) or live in extreme environments (such as Antarctica).
* Secondary Enrollees: Referred adult family members (such as siblings and spouses) of primary enrollees.
* Tertiary Enrollees: Adult persons from the general public can enroll to serve as matching controls. Tertiary enrollees will be screened based on age, gender, race and ethnicity, country of residence, disease/ conditions and employment history.
* Pregnant women may choose to enroll.

Exclusion Criteria:

* adults unable to consent,
* minors (under age 18)
* prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target population comprises of persons from many countries. Therefore, enrollees can be from other countries. However, biospecimen collection will occur in the USA.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2075-01-13 (Estimated); Study Completion 2075-01-13 (Estimated)

PRIMARY OUTCOMES:
Receipt of donated biospecimen for aerospace research | 50 years
  Donated biospecimens from participants will aid in the improvement of medical aerospace research. The key research divisions are cancer, cardiovascular, immunity and pathogenesis, neuroscience, and molecular microbiology.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Florida, Orlando, Florida, United States